CLINICAL TRIAL: NCT01409811
Title: A Pilot Study of the Impact of a Single Dose of Zoledronic Acid on Biomarkers in Breast Cancer
Brief Title: Biomarkers in Tissue Samples From Patients With Newly Diagnosed Breast Cancer Treated With Zoledronic Acid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed after it became too difficult to interest patients in participating.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10192; NCI-2011-02137 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Invasive Ductal Breast Carcinoma; Progesterone Receptor-positive Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (zoledronic acid) (Experimental): Patients receive a single dose of zoledronic acid 4 mg IV over 15 minutes on day 1. Patients then undergo planned definitive surgery (lumpectomy or mastectomy) on day 10-23. Tissue and blood samples from the initial biopsy and definitive surgery are collected to measure changes in biomarkers of tumor growth and metastasis, immunologic function, and the expression of genes important to breast cancer progression and metastasis.
  zoledronic acid: Given IV
  laboratory biomarker analysis: Correlative studies
  therapeutic conventional surgery: Undergo definitive lumpectomy or mastectomy
  Interventions: Drug: zoledronic acid; Other: laboratory biomarker analysis; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: zoledronic acid — Given IV
  Other Names: CGP 42446; CGP42446A; NDC-zoledronate; zoledronate; Zometa
Other: laboratory biomarker analysis — Correlative studies
Procedure: therapeutic conventional surgery — Undergo definitive lumpectomy or mastectomy

SUMMARY:
This pilot clinical trial studies biomarkers in tissue samples from patients with newly diagnosed breast cancer treated with zoledronic acid (ZA). Studying samples of tumor tissue in the laboratory from patients receiving ZA may help doctors learn more about the effects of ZA on cells. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate 14 tumor biomarkers of growth and metastasis (10 by microarray and 4 by RT-PCR) for change in response to ZA.

SECONDARY OBJECTIVES:

I. To evaluate 30 measures of immunologic function (by Luminex panel) for change in response to ZA a) after 48-72 hours and b) after 10-23 days.

II. To explore additional tumors biomarkers (approximately 20 by immunohistochemistry) for change in response to ZA.

OUTLINE: Patients receive zoledronic acid intravenously (IV) over 15 minutes on day 1. Patients then undergo planned definitive surgery (lumpectomy or mastectomy) on day 10-23. Tissue and blood samples from the initial biopsy and definitive surgery are collected to measure changes in biomarkers of tumor growth and metastasis, immunologic function, and the expression of genes important to breast cancer progression and metastasis.

After completion of study treatment, patients are followed up at 40-44 days.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Diagnosis of early stage, invasive ductal carcinoma (for which a lumpectomy or mastectomy is planned prior to systemic therapy)
* Estrogen receptor (ER)/progesterone receptor (PR) positive tumor (as confirmed by City of Hope Pathology Department if done on the outside) or
* Biopsy proven ER/PR positive tumor
* Ability to provide informed consent

Exclusion Criteria:

* Tumor that lacks both estrogen and progesterone receptors
* Patients who will receive neoadjuvant therapy prior to definitive surgery
* Bisphosphonate therapy currently or within the past 12 months
* Regular use of anti-inflammatory agents, with the exception of a baby aspirin regimen per principal investigator's (PI's) discretion
* Renal impairment as determined by a creatinine clearance < 60 ml/min as calculated by the Cockcroft-Gault formula using the patient's actual weight
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09-14; Primary Completion 2015-01-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Zoledronic Acid)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Insurance denial | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Zoledronic Acid)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 61 [50 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
  Hispanic | 2
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean (SE) Change From Pre-Treatment Baseline in (Log)pg/mL of Biomarker, by Time, Adjusted for Level at Baseline
Description: After the trial's premature closure, no data were collected for the primary endpoints; however, data on 14 of 30 secondary endpoints were obtained and are summarized below. Serum level (pg/mL) per biomarker was log-transformed. Change from baseline over time was evaluated using a generalized linear mixed model where follow-up time was represented by terms for the sequence of post-baseline samples or for (log)day on study. To recognize regression to the mean across repeated samples, a term for biomarker level at baseline, with or without interaction by time, was included when it improved the model's fit to the observed data. With 14 biomarkers sampled twice after baseline, there were 28 evaluations of change in biomarker level with exposure to study drug. Therefore, to control the False Discovery Rate (FDR), only evaluations that maintained the study's FDR at no more than 5 percent were accepted as true.
Time Frame: "48-72 hrs" and "Surgery (10-23 days)"
Population: The analysis included data from all evaluable subjects.
Measure: Mean (Standard Error); unit: (log)pg/mL
Arm/Group | Treatment (Zoledronic Acid)
Number analyzed (Participants) | 8
(log)pg/mL
  MIG @ 48-72 hrs | 2.31 (0.24)
  MIG @ Surgery (Day 10-23) | 0.62 (0.14)
  IP-10 @ 48-72 hrs | 1.47 (0.18)
  IP-10 @ Surgery (Day 10-23) | 0.16 (0.08)
  IL-12 @ 48-72 hrs | 0.23 (0.06)
  IL-12 @ Surgery (Day 10-23) | -0.01 (0.05)
  Eotaxin @ 48-72 hrs | -0.23 (0.06)
  Eotaxin @ Surgery (Day 10-23) | 0.02 (0.06)
  IL-2R @ 48-72 hrs | 0.17 (0.04)
  IL-2R @ Surgery (Day 10-23) | 0.10 (0.11)
  IFN-gamma @ 48-72 hrs | 0.04 (0.01)
  IFN-gamma @ Surgery (Day 10-23) | -0.01 (0.02)
  MIP1B @ 48-72 hrs | 0.37 (0.17)
  MIP1B @ Surgery (Day 10-23) | 0.28 (0.25)
  EGF @ 48-72 hrs | -0.18 (0.10)
  EGF @ Surgery (Day 10-23) | 0.25 (0.12)
  MCP-1 @ 48-72 hrs | 0.15 (0.08)
  MCP-1 @ Surgery (Day 10-23) | -0.02 (0.08)
  IFN-alpha per (log)Day until Surgery (Day 10-23) | -0.026 (0.000)
  MIP1A per (log)Day until Surgery (Day 10-23) | 0.12 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse events collected over a period of 2 years and 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Zoledronic Acid)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Zoledronic Acid) (N=9)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Pulmonary valve disease (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Tricuspid valve disease (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Eye infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Cholesterol high (Investigations) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Results shown come from the 8 evaluable subjects enrolled before early closure of the trial, originally planned to include 40 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes